CLINICAL TRIAL: NCT07035496
Title: The Effect of Benson's Relaxation Exercise on Anxiety and Kinesiophobia in Patients With Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Satı Danacı (Other)
Responsible Party: Sponsor-Investigator, Satı Danacı, Nurse, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-03/1181
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Total Knee Arthroplasty
Keywords: benson's relexation exercise; total knee arthroplasty; Kinesiophobia; anxiety
MeSH Terms: conditions — Kinesiophobia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 1. experimental group
  2. control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benson's Exercise Group (Experimental): Patients in the experimental group will be given an information brochure about the exercise by the researcher and the Benson Relaxation exercise will be explained. The patient will then perform the exercise under the control of the researcher. Then, the patient will be administered the exercise in the evening the day before surgery, in the morning of surgery, in the morning and evening on the 1st and 2nd postoperative days, and in the morning on the 3rd postoperative day. In addition to the Benson exercise, patients will receive routine treatment and care at the hospital.
  Interventions: Other: Benson's relaxation exercise
- Control group (No Intervention): patients will receive routine treatment and care at the hospital.

INTERVENTIONS:
Other: Benson's relaxation exercise — The Benson's relaxation exercise is based on the principle of choosing a word that is meaningful to the individual and focusing on it, breathing deeply and relaxing all the muscles in the body.The Benson relaxation exercise is a simple and easy-to-learn method.
  Arms: Benson's Exercise Group

SUMMARY:
The subject of the study is the effect of Benson Relaxation Exercise on anxiety and kinesiophobia in total knee arthroplasty patients.

DETAILED DESCRIPTION:
Sample of study was calculated using G*Power Software (ver. 3.1.9.2) for 95% power and medium effect size (f=0.40) at 95% confidence level i Participants were assigned to the experimental and control groups by block randomization method.

Patients in the experimental group will be given an information brochure about the exercise by the researcher and the Benson Relaxation exercise will be explained. The patient will then perform the exercise under the control of the researcher. Then, the patient will be administered the exercise in the evening the day before surgery, in the morning of surgery, in the morning and evening on the 1st and 2nd postoperative days, and in the morning on the 3rd postoperative day. In addition to the Benson exercise, patients will receive routine treatment and care at the hospital.

ELIGIBILITY:
* Patients 18-75 years of age
* Patients undergoing knee arthroplasty
* Patients who do not have communication problems, who are conscious and able to answer questions, and who do not have any disorder/disease affecting their decision-making ability (dementia, Alzheimer's, etc.)
* Patients who do not have psychiatric disorders such as anxiety disorder, panic attacks, depression and are not receiving psychiatric treatment such as antipsychotics/anxiolytics.
* Without Muscle Disease,
* Patients who volunteered to participate in the study.
* Patients who understand the study content and voluntarily sign the informed consent form for the study will be included in the study.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
The State Anxiety Scale | 1 day before surgery in the morning, half an hour before the surgery and 3 days postoperatively in the morning
  It is used to measure the level of anxiety. A minimum score of 0 and a maximum score of 80 can be obtained from the scale, and a high score indicates a high level of anxiety.
Tampa Kinesiophobia Scale | 1 day before surgery in the morning, half an hour before the surgery and 3 days postoperatively in the morning
  It is used to determine the level of kinesiophobia. While the minimum score value obtained from the scale is 17, the maximum score value is 68. A score above 37 on the scale is considered to be a high level of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Satı Danacı, Principal Investigator — Çankırı Public Hospital
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No